CLINICAL TRIAL: NCT04670549
Title: The Improve Osteoarthritis Care Study
Brief Title: Improve Osteoarthritis Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Nina Osteras, Senior researcher, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS 00203
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Implementation; Treatment guidelines
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre and post implementation phases (Other): Pre-implementation phase: during the pre-implementation period persons with hip or knee osteoarthritis will receive "usual care" as it is currently delivered by physiotherapists and general practitioners.
  Post-implementation phase: during the post-implementation phase patients with hip and knee OA will receive OA care more in line with the treatment recommendations.
  Interventions: Other: Implementation of treatment guidelines

INTERVENTIONS:
Other: Implementation of treatment guidelines — To improve knowledge of OA treatment recommendations among people with hip and knee OA, a lay language summary will be emailed all OA patient participants. A second summary of the treatment recommendations, targeting general practitioners (GPs) will also be emailed the OA patient participants. The patients will be encouraged to print and bring this summary to their GP at the next visit (user-initiated implementation). Barriers and facilitators for providing evidence-based OA care among primary care physiotherapists will be mapped through interviews. Thereafter, a tool-kit of strategies and practical aids intended to help overcome these barriers will be developed and made available for the physiotherapists.

SUMMARY:
The purpose of The Improve Osteoarthritis Care study is to improve the quality of osteoarthritis care in Norwegian primary care, by increasing the use of recommended treatment modalities and improving patient access to recommended treatments. The study will use tailored implementation strategies, targeting primary care physicians and physiotherapists to improve knowledge and addressing individual barriers to providing recommended treatments.

DETAILED DESCRIPTION:
Previous research has shown that current osteoarthritis care for persons with hip or knee osteoarthritis (OA) in Norway has a potential for improvement as the provided care may not necessarily reflect evidence-based guideline recommendations. The overall purpose of the "Improve Osteoarthritis Care" study is that people with symptomatic hip and knee OA should receive care in line with current recommendations. To achieve this goal, tailored implementation strategies will be applied in order to: 1) Improve the quality of care offered to people with symptomatic hip and knee OA, 2) increase knowledge of recommended OA care among people with hip and knee OA, 3) Increase the number of primary care physiotherapists' offering group-based patient-education and structured exercise as part of their routine clinical practice, 4) Increase the number of general practitioners who have received a summary of the OA treatment recommendations.

To evaluate the effect of the tailored implementation strategy a pre-post design will be applied, and members of the Norwegian Rheumatology Association with self-reported hip or knee OA will be asked to evaluate quality of OA care at the two timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported hip or knee osteoarthritis

Exclusion Criteria:

* Persons who do not understand the Norwegian language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1541 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The OsteoArthritis Quality Indicator questionnaire (OA-QI), version 2 | 18 months follow-up
  Assess change in patient-reported quality of OA care (mean total pass rate, 0-100 (best score))

CONTACTS AND LOCATIONS:
Overall Officials: Nina Østerås, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No